CLINICAL TRIAL: NCT06697197
Title: A Phase 1/2 Study of BMS-986482 as Monotherapy or Combination Therapy in Participants With Advanced Solid Tumors
Brief Title: A Study of BMS-986482 Alone or as Combination Therapy in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA236-0001; 2024-516602-28 (Other: EU CTR); U1111-1309-0886 (Other: WHO)
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
Keywords: Immuno-oncology; Regulatory T cells; Tregs
MeSH Terms: interventions — Nivolumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1A (Experimental)
  Interventions: Drug: BMS-986482
- Part 1B1 (Experimental)
  Interventions: Drug: BMS-986482; Drug: Nivolumab and rHuPH20
- Part 1B2 (Experimental)
  Interventions: Drug: BMS-986482; Drug: Nivolumab/relatlimab/rHuPH20
- Part 1B3 (Experimental)
  Interventions: Drug: BMS-986482; Drug: Bevacizumab
- Part 1C (Experimental)
  Interventions: Drug: BMS-986482
- Part 2A (Experimental)
  Interventions: Drug: BMS-986482
- Part 2B1 (Experimental)
  Interventions: Drug: BMS-986482; Drug: Nivolumab and rHuPH20
- Part 2B2 (Experimental)
  Interventions: Drug: BMS-986482; Drug: Nivolumab/relatlimab/rHuPH20
- Part 2B3 (Experimental)
  Interventions: Drug: BMS-986482; Drug: Bevacizumab

INTERVENTIONS:
Drug: BMS-986482 — Specified dose on specified days
Drug: Nivolumab and rHuPH20 — Specified dose on specified days
  Other Names: BMS-986298
  Arms: Part 1B1; Part 2B1
Drug: Nivolumab/relatlimab/rHuPH20 — Specified dose on specified days
  Other Names: BMS-986213
  Arms: Part 1B2; Part 2B2
Drug: Bevacizumab — Specified dose on specified days
  Arms: Part 1B3; Part 2B3

SUMMARY:
The purpose of this study is to test the safety and efficacy of BMS-986482 alone and as combination therapy in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* All participants must have a histologically or cytologically confirmed, advanced, unresectable/metastatic, solid malignancy measurable by RECIST v1.1, and have received, be refractory to, ineligible for, intolerant of, or refused existing therapy(ies) known to provide clinical benefit for the condition of the participant.
* Participant must be ≥ 18 years or the legal age of consent in the jurisdiction in which the study is taking place, inclusive, at the time of signing the ICF.

Exclusion Criteria:

* History of life threatening immune mediated toxicity related to prior T-cell agonist or checkpoint inhibitor therapy, except those that are unlikely to re-occur with standard countermeasures.
* Any significant acute or chronic medical illness which would interfere with study intervention or follow-up in the opinion of the investigator.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2029-01-04 (Estimated); Study Completion 2029-01-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) as assessed by National Cancer Institute -Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0) | Up to 135 days post last treatment visit
Number of participants with Serious AEs (SAEs) as assessed by NCI-CTCAE v5.0 | Up to 135 days post last treatment visit
Number of participants with AEs meeting protocol-defined Dose-Limiting Toxicity (DLT) criteria as assessed by NCI-CTCAE v5.0 | Up to Day 28
Number of participants with AEs leading to discontinuation as assessed by NCI-CTCAE v5.0 | Up to 135 days post last treatment visit
Number of deaths as assessed by NCI-CTCAE v5.0 | Through study completion (Up to 4 years)

SECONDARY OUTCOMES:
Concentration at the end of infusion (Cmax) | Up to 135 days post last treatment visit
Time of maximum observed concentration (Tmax) | Up to 135 days post last treatment visit
Area under the concentration-time curve in one dosing interval (AUC(TAU)) | Up to 135 days post last treatment visit
Overall Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) as assessed by Investigator | Up to 135 days post last treatment visit

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (21):
- United States (7):
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center, Irvine, California
  - The Angeles Clinic and Research Institute - West Los Angeles Office, Los Angeles, California
  - Local Institution - 0008, Aurora, Colorado
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Northwell Health/ RJ Zuckerberg Cancer Center, Lake Success, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Fred Hutchinson Cancer Center, Seattle, Washington
- UZ Gent, Ghent, Oost-Vlaanderen, Belgium
- Rigshospitalet, Copenhagen, Capital Region, Denmark
- France (2):
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Gustave Roussy, Villejuif, Paris
- Greece (2):
  - General Hospital of Athens "Laiko", Athens, Attikí
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki, Thessaloníki
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Milano
- Netherlands (2):
  - Nederlands Kanker Instituut Antoni van Leeuwenhoek (NKI AVL), Amsterdam, North Holland
  - Erasmus Medisch Centrum, Rotterdam
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario HM Sanchinarro, Madrid
- Karolinska Universitetssjukhuset Solna, Solna, Stockholms Län [se-01], Sweden

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06697197.html